CLINICAL TRIAL: NCT02249065
Title: MIRVASO® In Use Study: Managing Rosacea Through Assessment and Control of Its Erythema (The MIRACLE Study)
Brief Title: Mirvaso in Use Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.SPR.US 10305
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2017-11

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mirvaso Gel (Experimental): Brimonidine topical gel, 0.33%
  Interventions: Drug: Brimonidine

INTERVENTIONS:
Drug: Brimonidine
  Other Names: Mirvaso Gel

SUMMARY:
This study is designed to:

1. assess the signs and symptoms of rosacea, including erythema, without treatment and during treatment with Mirvaso® gel
2. further characterize lifestyle impact and patient satisfaction with Mirvaso® treatment
3. gain a better understanding of the real-world use of Mirvaso® on the pattern and management of facial erythema of rosacea.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years of age or older at time of study consent.
2. Subjects with a board certified dermatologist (BCD) clinical diagnosis of facial erythema of rosacea and eligible for treatment with Mirvaso® (brimonidine) topical gel, 0.33% per package insert.
3. Subjects with a clinician's erythema assessment (CEA) score of ~3 at Screening Visit 1.
4. Subjects with less than 3 facial inflammatory lesions of rosacea at Screening/Visit 1.
5. Subjects must be willing and able to give written informed consent including photography consent. Consent and photo consent will be obtained prior to any study related procedures
6. Females of childbearing potential with a negative urine pregnancy test (UPT) at Visit 1 (prior to test article application) or females of non-childbearing potential (deemed as post-menopausal [absence of menstrual bleeding for at least 1 year prior to enrollment], hysterectomy or bilateral oophorectomy).

Exclusion Criteria:

1. Subjects with particular forms of rosacea (rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin) or other concomitant facial dermatoses that are similar to rosacea such as peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus, or actinic telangiectasia.
2. Subjects with current diagnosis of Raynaud's syndrome, thromboangiitis obliterans, orthostatic hypotension, severe cardiovascular disease, cerebral or coronary insufficiency, renal or hepatic impairment, scleroderma, Sjogren's syndrome or depression.
3. Subjects with previous refractive eye surgery such as photorefractive keratectomy, laser-assisted sub-epithelial keratectomy, or laser-assisted in situ keratomileusis.
4. Current treatment with monoamine oxidase inhibitors.
5. Current treatment with barbiturates, opiates, sedatives, systemic anesthetics, or alpha- agonists.
6. Less than 3 months (90 days) stable dose treatment with tricyclic antidepressants, cardiac glycosides, beta blockers or other antihypertensive agents.
7. Subjects with any uncontrolled chronic or serious disease or medical condition that would normally prevent participation in a clinical study, or, in the judgment of the investigator, would put the subjects at undue risk, or might confound the study assessments (e.g., other dermatological diseases), or might interfere with the subjects' participation in the study, (e.g., planned hospitalization during the study).
8. Subjects who have received, applied, or taken treatments with drugs, cosmetics or devices known to cause facial erythema and who are deemed ineligible by the investigator.
9. Subjects with known allergies or sensitivities to any component of the study drug, including the active ingredient brimonidine tartrate label (refer to the package insert for Mirvaso® (brimonidine) topical gel, 0.33%).
10. Subjects with prior treatment with brimonidine gel, oxymetazoline or other (topical and/or systemic) alpha adrenergic agonists.
11. Subjects who are pregnant or breast-feeding or planning to become pregnant during the course of the study.
12. Subjects exposed to excessive ultraviolet (UV) radiation within I week prior to baseline and/or subject was unwilling to refrain from excessive exposure to UV radiation during the course of the study.
13. Subjects with the presence of a beard or excessive facial hair that would interfere with the study treatments or study assessments as deemed by the investigator, and refusal to remove beard or facial hair for duration of the study.
14. Subjects with non-stable dose of current (last 60 days) use of prescription rosacea medications.
15. Subjects with uncontrolled rosacea associated with inflammatory pustules and papules.
16. Study site staff, relatives of staff members, or other individuals who would have access to the clinical study protocol.
17. Subjects with participation in any investigational study within 30 days of entry into this study or concomitantly with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Sugarman, MD, Principal Investigator — Redwood Dermatology Center
Locations (12):
- United States (12):
  - Johnson Dermatology, Fort Smith, Arkansas
  - Blue Harbor Dermatology, Newport Beach, California
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - Redwood Dermatology Research, Santa Rosa, California
  - Florida Academic Dermatology Center, Miami, Florida
  - Research Institute of the Southeast, West Palm Beach, Florida
  - Grekin Skin Institute, Warren, Michigan
  - Advanced Skin Research Center, Omaha, Nebraska
  - Manhattan Dermatology and Cosmetic Surgery, New York, New York
  - DermDox Centers for Dermatology, Hazleton, Pennsylvania
  - Arlington Research Center, Arlington, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirvaso Gel: Brimonidine Gel (topical emulsion (gel), 0.33% brimonidine, once daily)
Period: Overall Study
Arm/Group | Mirvaso Gel
Started | 205
Treated | 181
Completed | 176
Not Completed | 29

BASELINE CHARACTERISTICS:
Population: ITT Population, Subjects who received at least 1 application of study drug, and completed at least 1 assessment
Groups:
- Mirvaso Gel: Brimonidine Gel
Arm/Group | Mirvaso Gel
Number analyzed (Participants) | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 143
  >=65 years | 38
Age, Continuous [Mean (Full Range); unit: years] | 52.4 [22.0 to 85.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 45
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 181

OUTCOME MEASURES:

1. Primary Outcome: Pre-Treatment Clinician Erythema Assessment (CEA)
Description: The number and percent of subjects in each CEA score category at each visit. CEA was conducted at the screening/baseline visit and all subsequent visits prior to the study drug application.
Time Frame: 14 days (Day 1 (Baseline), Day 7, and Day 14/Exit)
Population: Intent-to-treat (ITT) Population; Subjects who received at least 1 application of study drug, and completed at least 1 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Mirvaso Gel
Number analyzed (Participants) | 181
Participants
  Day 1 (Baseline): Clear Skin | 0
  Day 1 (Baseline): Almost Clear | 0
  Day 1 (Baseline): Mild Erythema | 7
  Day 1 (Baseline): Moderate Erythema | 144
  Day 1 (Baseline): Severe Erythema | 30
  Day 1 (Baseline): Missing | 0
  Day 7: Clear Skin | 3
  Day 7: Almost Clear | 18
  Day 7: Mild Erythema | 39
  Day 7: Moderate Erythema | 84
  Day 7: Severe Erythema | 24
  Day 7: Missing | 13
  Day 14: Clear Skin | 4
  Day 14: Almost Clear | 25
  Day 14: Mild Erythema | 39
  Day 14: Moderate Erythema | 86
  Day 14: Severe Erythema | 27
  Day 14: Missing | 0

2. Secondary Outcome: Subject Facial Redness Questionnaire
Description: Facial Redness Questionnaire at Day 1 and Day 14 (Mean Number of Subjects Who's Responses Indicate They Were/Were Not Bothered By Facial Redness, Across All 11 Facial Redness Questions)
Time Frame: 14 days (Day 1 (Baseline) and Day 14/Exit)
Population: ITT Population, Subjects who received at least 1 application of study drug, and completed at least 1 assessment
Measure: Mean (Standard Deviation); unit: Participants
Arm/Group | Mirvaso Gel
Number analyzed (Participants) | 181
Participants
  Not Bothered (Mean [SD], Day 1, Baseline) | 75.3 (39.4)
  Bothered (Mean [SD], Day 1, Baseline) | 104.7 (40.3)
  Missing (Day 1, Baseline) | 1 (0)
  Not Bothered (Mean [SD], Day 14) | 112.6 (28.9)
  Bothered (Mean [SD], Day 14) | 67.3 (26.2)
  Missing (Day 14) | 1.1 (.3)

3. Secondary Outcome: Subject Treatment Satisfaction Questionnaire
Description: Mean Subject Treatment Satisfaction at Day 14 (Average Response Across 12 Questions)
Time Frame: 14 days (Day 14/Exit)
Population: ITT Population, Subjects who received at least 1 application of study drug, and completed at least 1 assessment
Measure: Mean (Standard Deviation); unit: Participants
Arm/Group | Mirvaso Gel
Number analyzed (Participants) | 181
Participants
  Satisfied Participants (Mean [SD]) | 127.3 (22.2)
  Dissatisfied Participants (Mean [SD]) | 52.7 (22.2)
  Missing | 1.0 (0.0)

4. Secondary Outcome: Facial Redness Visual Analog Scale (VAS)
Description: The number and percent of subjects in each transformed response category for the in-office subject reported facial redness VAS
Time Frame: 14 days (Day 1 (Baseline), Day 14/Exit)
Population: ITT Population, Subjects who received at least 1 application of study drug, and completed at least 1 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Mirvaso Gel
Number analyzed (Participants) | 181
Participants
  Day 1: None | 1
  Day 1: Very Mild | 31
  Day 1: Mild | 57
  Day 1: Moderate | 48
  Day 1: Severe | 38
  Day 1: Very Severe | 6
  Day 14: None | 1
  Day 14: Very Mild | 63
  Day 14: Mild | 45
  Day 14: Moderate | 44
  Day 14: Severe | 22
  Day 14: Very Severe | 6

5. Secondary Outcome: Inflammatory Lesions
Description: Change from baseline in facial inflammatory lesion count
Time Frame: 14 days (Day 1 (Baseline) and Day 14/Exit)
Population: ITT Population, Subjects who received at least 1 application of study drug, and completed at least 1 assessment
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Mirvaso Gel
Number analyzed (Participants) | 181
lesions
  Day 1: Lesions | .6 (1.2)
  Day 14: Lesions | 1.5 (4.4)
  Day 14: Change From Baseline | 1 (3.9)

ADVERSE EVENTS:
Time Frame: 29 Days
Description: Adverse events were recorded for at least 14 days prior to the first treatment application.
Arm/Group | Mirvaso Gel
Serious Adverse Events (participants affected / at risk) | 3/181
Other Adverse Events (participants affected / at risk) | 68/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirvaso Gel (N=181)
myocardial infarction (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mirvaso Gel (N=181)
condition aggravated (General disorders) | 33
feeling hot (General disorders) | 4
rosacea (Skin and subcutaneous tissue disorders) | 21
Erythema (Skin and subcutaneous tissue disorders) | 7
nasopharyngitis (Infections and infestations) | 6

LIMITATIONS AND CAVEATS:
Open label, single arm, short duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days